CLINICAL TRIAL: NCT05062161
Title: Nocturnal Hypertension and Sleep (Sleep BP Study)
Brief Title: Sleep Duration and Blood Pressure During Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Marwah Abdalla, Associate Professor of Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AAAT8157; K23HL141682-01 (NIH)
Record Dates: First submitted 2021-09-24; First posted 2021-09-30 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Blood Pressure; Hypertension; Elevated Blood Pressure; Sleep; Short Sleep Phenotype
Keywords: Nocturnal Hypertension; Short Sleep Duration; Cardiovascular Disease
MeSH Terms: conditions — Hypertension; Sleep Wake Disorders; Cardiovascular Diseases | interventions — sodium bicarbonate-based toothpaste

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will be randomized in a 1:1 ratio to each arm by a computer-generated random allocation sequence. All study investigators and outcome assessors will be blinded to group assignment and will not have access to the randomization sequence. The Educational Research Coordinator who will deliver the educational sessions will be unblinded to treatment arm but will not be involved in collecting study measures or data analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Hygiene/Extension Intervention (Experimental): Participants with short sleep duration will receive a 60-minute educational session on sleep hygiene/extension. Over an 8-week period, participants will receive weekly phone or Zoom video calls from the Educational Research Coordinator to review additional materials including handouts and/or complete questionnaires about sleep. Participants will undergo sleep tracking/monitoring during the 8-week period, and repeat BP/heart rate monitoring for 24 hours after the 8-week period.
  Interventions: Behavioral: Sleep hygiene/extension intervention
- Control Condition (Active Comparator): Participants with short sleep duration will receive a 60-minute educational session on sleep physiology. Over an 8-week period, participants will receive weekly phone or Zoom video calls from the Educational Research Coordinator to review additional materials including handouts. Participants will undergo sleep tracking/monitoring during the 8-week period, and repeat BP/heart rate monitoring for 24 hours after the 8-week period.
  Interventions: Behavioral: Control care

INTERVENTIONS:
Behavioral: Sleep hygiene/extension intervention — The 60-minute sleep hygiene/extension educational session include the following: This session will consist of questionnaires, handouts, videos, and a discussion. Topic examples include information on establishing a comfortable sleep environment, including strategies on how to extend sleep duration by a maximum of 1 hour over the duration of the 8-week trial for an average of 7.5 minutes per week, not to exceed 15 minutes per week. Participants will also receive educational brochures and a sleep diary.
  Arms: Sleep Hygiene/Extension Intervention
Behavioral: Control care — The 60-minute educational session will address sleep physiology but not sleep hygiene. This session will consist of questionnaires, handouts, videos, and a discussion. Participants will receive an educational brochure.
  Arms: Control Condition

SUMMARY:
The purpose of this study is to examine the impact that sleep duration has on blood pressure (BP) levels during sleep. The investigator will examine the effect of an 8-week sleep hygiene/extension intervention vs. control on sleep BP.

DETAILED DESCRIPTION:
Short sleep duration (SSD), defined as sleeping less than 7 hours per night, affects over 33% of US adults and is associated with increased mortality. SSD is a modifiable risk factor for obesity, type 2 diabetes, and HTN. Cross-sectional studies have demonstrated that SSD is associated with higher sleep BP levels. SSD is also associated with non-dipping BP which is primarily explained by higher sleep BP levels. However, many of the cross-sectional studies have included adolescent participants or have not used reference standard measures of sleep duration such as wrist actigraphy. Manipulating sleep duration experimentally through sleep restriction or deprivation is associated with higher 24-hour and sleep BP levels. In contrast, there is scarce data on the effect of sleep extension on sleep BP levels among adults with SSD.

Eligible community individuals with short sleep duration will be randomized to sleep extension vs. control using 24-hour ambulatory blood pressure monitoring (ABPM) and actigraphy in the naturalistic environment. Individuals will be assessed throughout the study using questionnaires, activity monitoring via a Fitbit device (for 8 weeks), blood pressure monitoring using a 24-hour ABPM device, and heart rate variability monitoring for 24-hours.

ELIGIBILITY:
Inclusion Criteria:

* English speaking adults
* Age 18 and older
* Sleep duration < 7 hours per night as assessed via daily self-report of sleep hours

Exclusion Criteria:

* Inability to read or write in English
* Pregnant or plans to get pregnant within study period
* Arm circumference >50 cm
* Lymphedema of the arm or unable to wear ABPM device for 24 hours or wrist actigraphy for 8 weeks
* End-stage renal disease (ESRD) on dialysis
* Unreliable internet or phone/text access
* High risk of Obstructive Sleep Apnea (OSA) (using the Berlin Questionnaire or diagnosis of OSA or use continuous positive airway pressure device)
* High risk of insomnia (using the Insomnia Severity Index), or a known prior history of insomnia, and/or use of prescription sleep aides
* High risk of depression (using the Patient Health Questionnaire Depression Scale: PHQ-8)
* Perimenopausal women who have hot flashes (using the Menopause Rating Scale (MRS) questionnaire, administered only to females age 45-65)
* Plan to travel out of state and/or internationally during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marwah Abdalla, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University Center for Behavioral Cardiovascular Health: CBCH, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 66 participants enrolled in the study. 1 participant withdrew prior to randomization.
Period: Overall Study
Arm/Group | Sleep Hygiene/Extension Intervention | Control Condition
Started | 32 | 33
Completed | 32 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Condition | Sleep Hygiene/Extension Intervention | Total
Number analyzed (Participants) | 33 | 32 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (16.6) | 36.7 (15.1) | 37.3 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 14 | 13 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 7 | 17
  Not Hispanic or Latino | 23 | 24 | 47
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 11 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 7 | 15
  White | 10 | 9 | 19
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 33 | 32 | 65

OUTCOME MEASURES:

1. Primary Outcome: Mean Sleep Systolic Blood Pressure (BP) at Baseline and 8 Weeks
Description: Mean of valid BP readings during the sleep period on 24-hour ambulatory blood pressure monitor will be calculated to obtain mean sleep systolic BP (mmHg) at baseline and 8 weeks.
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Control Condition | Sleep Hygiene/Extension Intervention
Number analyzed (Participants) | 33 | 32
mmHg
  Baseline | 100.8 (13.3) | 100.0 (9.1)
  8 Weeks | 101.4 (13.2) | 102.3 (12.7)

2. Primary Outcome: Mean Sleep Diastolic Blood Pressure (BP) at Baseline and 8 Weeks
Description: Mean of valid BP readings during the sleep period on 24-hour ambulatory blood pressure monitor will be calculated to obtain mean sleep diastolic BP (mmHg) at baseline and 8 weeks.
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Control Condition | Sleep Hygiene/Extension Intervention
Number analyzed (Participants) | 33 | 32
mmHg
  Baseline | 58.6 (8.2) | 57.9 (6.5)
  8 weeks | 60.0 (7.8) | 60.1 (6.4)

3. Secondary Outcome: Mean Awake Systolic Blood Pressure (BP) at Baseline and 8 Weeks
Description: Mean of valid BP readings during the awake period on 24-hour ambulatory blood pressure monitor will be calculated to obtain mean awake systolic BP (mmHg) at baseline and 8 weeks.
Time Frame: Baseline, 8 weeks
Reporting Status: Not Posted, anticipated posting 2025-12

4. Secondary Outcome: Mean Awake Diastolic Blood Pressure (BP) at Baseline and 8 Weeks
Description: Mean of valid BP readings during the awake period on 24-hour ambulatory blood pressure monitor will be calculated to obtain mean awake diastolic BP (mmHg) at baseline and 8 weeks.
Time Frame: Baseline, 8 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Mean 24-hour Systolic Blood Pressure (BP) at Baseline and 8 Weeks
Description: Mean of valid BP readings during the awake period on 24-hour ambulatory blood pressure monitor will be calculated to obtain mean awake 24-hour systolic BP (mmHg) at baseline and 8 weeks.
Time Frame: Baseline, 8 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Mean 24-hour Diastolic Blood Pressure (BP) at Baseline and 8 Weeks
Description: Mean of valid BP readings during the awake period on 24-hour ambulatory blood pressure monitor will be calculated to obtain mean awake 24-hour diastolic BP (mmHg) at baseline and 8 weeks.
Time Frame: Baseline, 8 weeks
Reporting Status: Not Posted

7. Secondary Outcome: 24-hour High Frequency Heart Rate Variability
Description: 24-hour high frequency heart rate variability will be estimated from R-R interval data from the Cardio SOLO device at baseline and 8 weeks and compared across randomization arms.
Time Frame: Baseline, 8 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Actigraphy-derived Mean Sleep Duration
Description: This is to measure if the intervention (sleep hygiene/extension) would increase mean sleep duration for participants randomized to sleep hygiene/extension, actigraphy-derived sleep duration will be used to evaluate the intervention. Actigraphy-derived mean sleep duration will be calculated daily as the total time between the sleep and awake period as defined on the Fitbit device in number of hours.
Time Frame: 8 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Control Condition | Sleep Hygiene/Extension Intervention
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/32
Other Adverse Events (participants affected / at risk) | 0/33 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-11): https://cdn.clinicaltrials.gov/large-docs/61/NCT05062161/Prot_SAP_000.pdf